CLINICAL TRIAL: NCT05101005
Title: A Prospective, Multi-center, Randomized Trial Comparing the Long-term Efficacy of Drug-coated Balloon Versus Drug-eluting Stent in Large de Novo Coronary Lesions
Brief Title: Long-term Efficacy of Drug-coated Balloon Versus Drug-eluting Stent in Large de Novo Coronary Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJDCB-01
Record Dates: First submitted 2021-10-13; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease; Drug-coated Balloon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-coated balloon (Experimental): Drug-coated balloon is used to treat coronary artery stenosis lesions and improve myocardial blood flow.
  Interventions: Device: Drug-Coated Balloon
- Sirolimus-Eluting Stent (Active Comparator): Sirolimus-Eluting Stent is treated for coronary artery stenosis lesions.
  Interventions: Device: Sirolimus-Eluting Stent

INTERVENTIONS:
Device: Drug-Coated Balloon — Drug-coated balloon is a fast-exchange balloon dilatation catheter, used to treat coronary artery stenosis lesions.
  Arms: Drug-coated balloon
Device: Sirolimus-Eluting Stent — Sirolimus-Eluting Stent is treated for coronary artery stenosis lesions.
  Arms: Sirolimus-Eluting Stent

SUMMARY:
To evaluate the efficacy of drug-coated balloon versus drug-eluting stent for the treatment of large de novo coronary lesions(RVD=2.75~4.0mm).

DETAILED DESCRIPTION:
Patients were randomly assigned (1:1) to receive angioplasty with DCB or implantation of a DES. Dual anti-platelet therapy was given according to current guidelines. Follow-up was originally scheduled at by telephone or clinical visit at 1 month, 6 months, and 12 months after discharge. The primary endpoint is a composite endpoint of cardiac death, target vessel related myocardial infarction, and target lesion revascularization (TLF) at 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤80 years, regardless of gender;
2. De novo lesion in a native coronary artery;
3. Stable angina, or unstable angina, or old myocardial infarction or asymptomatic myocardial ischemia;
4. Reference vessel diameter is 2.75mm-4.0mm with diameter stenosis ≥70% or ≥50% (with evidence of ischemia) and TIMI flow ≥1;
5. The subject can receive any type of coronary vascular revascularization (including balloon angioplasty, stent implantation or coronary artery bypass grafting);
6. The subject who can understand the purpose of the trial, voluntarily participate in and sign an informed consent form, and is willing to accept clinical follow-up.

Exclusion Criteria:

1. Reference vessel diameter <2.75 mm or >4.0 mm;
2. In stent restenosis;
3. Left main lesion, chronic complete occlusion lesion;
4. Ostial lesion ≤2mm from the LM, or bifurcation lesion with branch vessel diameter≥2.5mm;
5. There is a large scale of thrombus in the target vessel, and the thrombus grade >3 after thrombolysis or aspiration;
6. Severe heart failure (NYHA IV);
7. Severe renal failure (GFR<30ml/min) or undergoing hemodialysis treatment;
8. Severe liver failure (bilirubin is over 2 times the upper limit of normal, or alanine aminotransferase is over 3 times the upper limit of normal);
9. Patients with vein graft restenosis after bypass or severe heart valve disease;
10. Pregnant or breastfeeding female patients;
11. The life expectancy of the patient is less than 12 months;
12. The subject cannot be treated with anticoagulation because of bleeding tendency, history of active peptic ulcer, stroke in the 6 months before surgery, anti-platelet agents or anticoagulant treatment contraindications;
13. Anemia (women's hemoglobin <117g/L, or men's hemoglobin <134g/L), or thrombocytopenia detected before the intervention within 6 months (<100×10⁹/L);
14. Planned to perform non-cardiac surgery within 12 months after index procedure;
15. The subject who participated in other clinical trials of drugs or instruments and did not reach time of primary endpoint;
16. Heart transplant patients;
17. Allergic to aspirin, clopidogrel, heparin, contrast agents, or paclitaxel;
18. The investigator judged that the patient had poor compliance and could not complete the study as required.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure | 12 months follow-up
  A composite endpoint consisting of cardiac death, target vessel-related myocardial infarction, and target lesion revascularization

SECONDARY OUTCOMES:
Procedural success | During the hospital stay, up to 7 days after PCI
  Consisting of device success ( after successful delivery of the study balloon, the visual residual stenosis of the target lesion is less than 50%, TIMI level 3 blood flow ) , Lesion success (defined as the proportion of the target lesions in which the final stenosis is <20% after treatment with any other adjunctive therapy ) , Clinical success ( Defined as no major adverse cardiac events caused by ischemia during the subject's hospitalization).
Target lesion failure | 1 month, 6months follow-up
  A composite endpoint consisting of cardiac death, target vessel-related myocardial infarction, and target lesion revascularization
Patient-oriented composite endpoint | 1 month, 6months,12 months follow-up
  A composite of all-cause mortality, myocardial infarction, and any revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Yansong Li, Principal Investigator — Shanghai Songjiang Central Hospital

IPD SHARING:
Plan to Share IPD: No